CLINICAL TRIAL: NCT05824533
Title: Difference in Patellar Tracking Before and After Journey II BCS Total Knee Arthroplasty, Evaluated With 4D CT Imaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to financial constraints, the study could not be continuedout as planned. Enrolled participants will finish treatment per study protocol.
Sponsor: Sebastiaan van de Groes (Other)
Collaborators: Smith & Nephew, Inc. (Industry); Treant, the Netherlands (Unknown)
Responsible Party: Sponsor-Investigator, Sebastiaan van de Groes, Principal investigator & Orthopeadic surgeon, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4DCT-tracking-TKA
Record Dates: First submitted 2023-03-22; First posted 2023-04-21 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Knee; Replacement; Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TKA with onlay patella button (Experimental): Total knee arthroplasty (TKA) with a patella placed with the use of the CORI based on pre-operative 4DCT images of the knee.
  Interventions: Device: onlay patella button
- TKA without onlay patella button (Active Comparator): Total knee arthroplasty (TKA) placed with the use of the CORI based on pre-operative 4DCT images of the knee.
  Interventions: Procedure: Conventional procedure; NO onlay patella button

INTERVENTIONS:
Device: onlay patella button — Total knee arthroplasty (TKA) with a patella onlay button placed with a CORI Robotics System based on pre-operative 4DCT-imaging.
  Arms: TKA with onlay patella button
Procedure: Conventional procedure; NO onlay patella button — Total knee arthroplasty (TKA) placed with a CORI Robotics System based on pre-operative 4DCT-imaging.
  Arms: TKA without onlay patella button

SUMMARY:
The current proposal aims to investigate the patellar tracking in adult patients receiving Journey II Bi-Cruciate Stabilized (BCS) total knee arthroplasty (TKA) before and one year after surgery, positioned with the CORI Robotics System instrumentation. The hypothesis is that less change in patella tracking before and after surgery will lead to less anterior knee pain complaints. Patella tracking is investigated using 4Dimensional Computer Tomography (4D CT) imaging.

Researchers will compare the group of participants that will receive a patella onlay button with the group that will not receive a patella onlay button with their TKA to see if there is a difference in motion and pain experienced by the participants.

DETAILED DESCRIPTION:
Rationale: Pain at the anterior side of the knee after total knee arthroplasty is still a common phenomenon with an incidence reported to be as high as 49 percent. The aetiology is poorly understood and several mechanisms have been postulated. Next to the influence of alignment on retinacular stresses, overstuffing of the patellofemoral joint and instability also lead to higher retinacular stresses and are shown to lead to anterior knee pain. These mechanisms are all related to surgical technique and implant positioning. There are also mechanisms related to prosthesis design, like the sagittal curve, trochlear depth and trochlea shape.

New implant designs like the Journey II prothesis are designed to replicate optimal geometry and optimal tibiofemoral and patellofemoral kinematics. Therefore, the Journey II Bi-Cruciate Stabilized (BCS) seems the optimal implant to reduce anterior knee pain. However, large registry studies show that a higher revision rate is seen when no patellar button is used in case of the Journey II BCS. The use of a patellar button is still under debate, but using an onlay patella button has clear influence on the patella tracking. Therefore, there might be a relation between the use of an onlay patella button and the retinacular balance and thus clinical results.

With current surgical instrumentation the positioning of the prosthesis based on the kinematics of the natural knee is challenging, and a small error can completely counteract the normal motion defined by the implant design/geometry. Therefore, comparative studies are only leading to new evidence when the surgical technique is including objective and accurate tools, like the CORI robotic platform. With the CORI, component positioning can be set based on constitutional alignment and ligament functioning. Furthermore, the patellofemoral compartment can be taken into account during the surgery to enable optimal geometry replication of the trochlea in the sagittal plane. This enables the surgeon to position the components accurately within the envelop of motion of a specific joint.

With new emerging imaging techniques, the investigators are able to investigate in vivo patella tracking. One of these promising techniques is the 4D CT imaging. This technique is proven to be accurate within 1 mm and 1° and therefore useful to investigate the patellofemoral compartment.

The current proposal aims to investigate the patellar tracking in patients receiving Journey II BCS total knee arthroplasty (TKA) before and one year after surgery, positioned with the CORI Robotics System instrumentation. The hypothesis is that less change in patella tracking before and after surgery will lead to less anterior knee pain complaints. Patella tracking is investigated using 4Dimensional Computer Tomography (4D CT) imaging.

Research participants/locations:

A total of 100 participants will be included in the study from two sites in the Netherlands (Radboudumc and Treant medical centers). Half of the participants will undergo TKA placed with the CORI Robotics and a patella onlay button and the other half (50 participants) will undergo a TKA placed with the CORI Robotics System and without a patella onlay button.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory knee osteoarthritis, which is confirmed by radiology.
* Osteoarthritis is unilateral or bilateral with the contralateral knee functioning properly, not operated on in the last 6 months.
* Set to receive a primary cemented total knee arthroplasty.
* Aged between 50 and 80 years, inclusive, on the day of the operation.

  * This age limit of 50 is based on the desire to include exclusively patients with primary osteoarthritis. As osteoarthritis is an age-related disorder, it generally involves adults over the age of 50 years. Patients under the age of 50 years who present with osteoarthritis usually have osteoarthritis due to a secondary cause (e.g. post-traumatic osteoarthritis).
  * A maximum age of 80 years will be employed. This age limit will be adopted because patients should be well able to perform an extension-flexion movement while a dynamic CT scan is made.
* In stable health (American Society of Anesthesiology (ASA)-score ≤ 3) and is free of or treated for cardiac, pulmonary, haematological, or other conditions that would pose excessive operative risk.
* Patient has a correctable or <10° rigid (non-correctable) varus deformity of the knee.
* Participants must be able to give informed consent.
* Patient plans to be available for follow-up until two years post-operative.
* Ability to walk for 2 minutes without walking aid

Exclusion Criteria:

* Valgus deformity
* Body MAss Index (BMI) > 35.
* Previous hip /knee/ankle replacement surgery in the last 12 months, or is planned to have a hip replacement in the next 6-12 months.
* Patient has had major, non-arthroscopic surgery to the study knee, including High Tibial Osteotomy (HTO).
* Patient has an active, local infection or systemic infection
* Incomplete or insufficient tissue surrounding the knee.
* Severe damage to the medial or collateral knee ligaments and popliteal tendon
* Documented osteoporosis with patient in active medical treatment.
* Patient has physical, emotional or neurological conditions that impacts gait or balance, or would compromise compliance with post-operative rehabilitation and follow-up.
* Bone quality compromised by disease or infection which cannot provide adequate support and/or fixation to the prosthesis
* Knee flexion < 90 degrees
* > 30 degrees extension deficit (active restraint to extension)
* Patient does not have a proper functioning patella tendon on the affected side; measured as inability of active extension of the knee
* Patient has active rheumatoid arthritis, any auto-immune disorder, immunosuppressive disorder or a terminal illness.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Changes in patellar shift during knee flexion between the pre- and one year post-operative situation | pre-operative, and 12 months post-operative
  This will be measured with 4DCT imaging.
Changes in patellar tilt during knee flexion between the pre- and one year post-operative situation | pre-operative, and 12 months post-operative
  This will be measured with 4DCT imaging.
Difference between pre-operative and one year post-operative in pain | pre-operative, and 12 months post-operative
  Pain will be measured using the NRS scale. The numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.
Difference in patella tracking between patients with and without an onlay patella button | pre-operative, and 12 months post-operative
  This will be measured with 4DCT imaging. The Patellar Center - Trochlear Groove distance will be used to quantify patellar tracking throughout an extension-flexion movement.

SECONDARY OUTCOMES:
Implant positioning | during surgery
  By using the CORI, the investigators will collect implant position.
Patient Reported Outcome Measures (PROMs): Forgotten Joint Score (FJS) | pre-operative, 3, 6, 12 months post-operative
  Forgotten Joint Score (FJS). To assess joint-specific patient reported outcomes in TKA participants. Responses to 12 questions are recorded with a five point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale and then reversed with a high value reflecting the ability of the participant to forget about the replaced knee joint during the activities of daily living. A score of 100 is the best possible outcome.
PROMs: Knee Injury and Osteoarthritis Outcome Score (KOOS) | pre-operative, 3, 6, 12 months post-operative
  Knee Injury and Osteoarthritis Outcome Score (KOOS): Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
PROMs: Kujala knee score | pre-operative, 3, 6, 12 months post-operative
  To assess participiant experienced outcomes in pain and movement before and after the TKA
PROMs: EuroQol Five-Dimensional Five-Level (EQ-5D-L) | pre-operative, 3, 6, 12 months post-operative
  To assess the participant's health state in TKA participants. The EQ-5D-5L is composed of the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the five dimensions are combined in a 5-digit code. The EQ- 5D-5L index value is derived by using the vendor supplied calculator to convert each 5-digit EQ-5D-5L profile. The EQ VAS corresponds to a 20 cm vertical, visual analogue scale ranging from 'the best health you can imagine' to 'the worst health you can imagine'. A higher number is a better outcome.
PROMs: Numeric Rating Scale (NRS) | pre-operative, 3, 6, 12 months post-operative
  The numeric rating scale (NRS) is a pain screening tool, used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiaan van de Groes, MD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Treant, the Netherlands, Groningen
  - RadboudUMC, Nijmegen